CLINICAL TRIAL: NCT06758583
Title: An Open-label, Randomized, Parallel-group, Single-center Trial to Compare Pharmacokinetics of Dapiglutide After a Single Subcutaneous Dose of the Drug Product Concentrations 10 mg/mL or 25 mg/mL in Participants With Overweight or Obesity
Brief Title: A Trial Comparing Pharmacokinetics, Safety and Tolerability of Two Subcutaneous Concentrations of Dapiglutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZP7570-24026; 2024-516901-21 (EudraCT Number)
Record Dates: First submitted 2024-12-09; First posted 2025-01-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obesity
Keywords: GLP-1R/GLP-2RA; overweight; obesity; weight management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This is a phase 1, open-label, single-center, randomized, parallel-group trial designed to investigate the pharmacokinetic profiles, safety, and tolerability of a single dose administration of 7.5 mg dapiglutide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapiglutide 10 mg/mL (Experimental): Single dose, s.c. administration
  Interventions: Drug: Dapiglutide 7.5 mg
- Dapiglutide 25 mg/mL (Experimental): Single dose, s.c. administration
  Interventions: Drug: Dapiglutide 7.5 mg

INTERVENTIONS:
Drug: Dapiglutide 7.5 mg — Single dose administration of 7.5 mg dapiglutide administered s.c. with two drug product concentrations, 10 mg/mL and 25 mg/mL.

SUMMARY:
This is a phase 1, open-label, single-center, randomized, parallel-group trial designed to investigate the pharmacokinetic profiles, safety, and tolerability of a single dose administration of 7.5 mg dapiglutide administered s.c. with two drug product concentrations, 10 mg/mL and 25 mg/mL. The trial will be conducted in participants with a BMI ≥ 27.0 kg/m2.

DETAILED DESCRIPTION:
Dapiglutide is a dual Glucagon-like peptide-1-/Glucagon-like peptide-2 Receptor Agonist (GLP-1R/GLP-2RA) in clinical development for weight management. The purpose of this phase 1 trial is to compare pharmacokinetics (PK) of a single dose administration of 7.5 mg dapiglutide administered subcutaneously (s.c.) with two drug product concentrations, 10 mg/mL and 25 mg/mL and will be conducted in 30 participants with a body mass index (BMI) ≥ 27.0 kg/m2. The development of a drug product with higher drug concentration will facilitate investigation of a wider dose range of dapiglutide in the clinical development program of the compound. The PK profile of a weight management drug should be assessed in people with a wide range of BMI and with a BMI within the range of the target population as body weight is expected to influence PKs of dapiglutide.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 64 years, both inclusive,
* BMI >= 27.0 kg/m^2
* HbA1c < 6.5 %.

Exclusion Criteria:

* Any history or presence of a disorder or a disease, which, in the investigator's opinion, might jeopardize participant's safety, evaluation of results or compliance with the protocol, treatment with dapiglutide (any exposure) or any other drugs, including dual and tri agonists, involving a GLP-1 RA or GLP-2 RA within 180 days prior to screening.
* Any medication (prescription and non-prescription drugs) with the exception of stable treatment with antihypertensive and lipid-lowering drugs as well as thyroid replacement therapy.
* Female participants of childbearing potential who are not willing to use highly effective contraception until 42 days after dosing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants of childbearing potential who are not willing to use highly effective contraception until 42 days after dosing are not eligible to participate
Enrollment: 30 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
To compare pharmacokinetics of a single dose administration of 7.5 mg dapiglutide | Trial Day 1 to 28
  Area under the dapiglutide plasma concentration-time curve from time zero to infinity after a single 7.5 mg dose of dapiglutide (AUC0-inf).
To compare pharmacokinetics of a single dose administration of 7.5 mg dapiglutide | Trial Day 1 to 28
  Maximum observed dapiglutide plasma concentration after a single 7.5 mg dose of dapiglutide (Cmax)

SECONDARY OUTCOMES:
To characterize the pharmacokinetic profiles of a single dose administration of 7.5 mg dapiglutide | Day 1 to 28
  Area under the dapiglutide plasma concentration-time curve from time zero to last measurable concentration after a single 7.5 mg dose of dapiglutide (AUC0-t)
To characterize the pharmacokinetic profiles of a single dose administration of 7.5 mg dapiglutide | Day 1 to 28
  Time to maximum observed dapiglutide plasma concentration after a single 7.5 mg dose of dapiglutide (Tmax)
To characterize the pharmacokinetic profiles of a single dose administration of 7.5 mg dapiglutide | Day 1 to 28
  Terminal elimination half-life for dapiglutide after a single 7.5 mg dose of dapiglutide (t½)
To characterize the pharmacokinetic profiles of a single dose administration of 7.5 mg dapiglutide | Day 1 to 28
  Elimination rate constant for dapiglutide after a single 7.5 mg dose of dapiglutide (λz)
To characterize the pharmacokinetic profiles of a single dose administration of 7.5 mg dapiglutide | Day 1 to 28
  Apparent clearance of dapiglutide after a single 7.5 mg dose of dapiglutide (CL/F)
To characterize the pharmacokinetic profiles of a single dose administration of 7.5 mg dapiglutide | Day 1 to 28
  Apparent volume of distribution during terminal phase of dapiglutide after a single 7.5 mg dose of dapiglutide (Vz/f)
To characterize the pharmacokinetic profiles of a single dose administration of 7.5 mg dapiglutide | Day 1 to 28
  Mean residence time of dapiglutide after a single 7.5 mg dose of dapiglutide (MRT)
To investigate the safety and tolerability of a single dose administration of 7.5 mg dapiglutide | Day 1 to 42
  Incidence of treatment emergent adverse events (TEAEs) from dosing (Day 1) to end of trial (Day 42).

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hoevelmann, MD, Principal Investigator — Profil, Neuss
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
The data collection and handling of clinical trial data at the trial site has been designed to limit the possibility of identifying trial subjects from their data. To this end, pseudonymised data will be used wherever possible and the collection of demographic information that could be used for re-identification of subjects will be restricted to the extent necessary for the conduct of this trial.